CLINICAL TRIAL: NCT01714921
Title: ProSA Protecta Smart Analysis Register
Brief Title: Protecta Smart Analysis Register
Acronym: ProSA
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic GmbH Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: CEN_G_CA_13
Record Dates: First submitted 2012-10-16; First posted 2012-10-26 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2018-04

CONDITIONS: Patients With an Indication for an ICD Implantation According to the Guidelines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICD patients: Patients with an indication for an ICD implantation according to the guidelines treated with a Protecta™, Protecta™ XT or any equivalent following product

SUMMARY:
ProSA is a prospective, non-randomized, multicenter, observational study investigating the utilization and effectiveness of the Smart Shock™ algorithm in ICD patients treated with a Protecta™, Protecta™ XT or any equivalent following product.

ELIGIBILITY:
Inclusion Criteria:

* patients implanted with an Implantable Cardioverter Defibrillator (ICD) with the smart shock algorithm (Protecta™, Protecta™ XT or any equivalent following product)
* written informed consent

Exclusion Criteria:

* patients with life expectancy less than 24 months
* patients younger than 18 years
* pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that satisfy the inclusion criteria and signed the informed consent
Sampling Method: Non-Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2010-06-09 (Actual); Primary Completion 2015-01-05 (Actual); Study Completion 2015-01-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 504 patients were enrolled at 29 German sites between 09-Jun-2010 and 22-Oct-2012
Groups:
- ICD Patients (Single Arm Study): Patients with an indication for an Implantable Cardioverter/Defibrillator (ICD) implantation according to the guidelines treated with a Protecta™, Protecta™ XT or any equivalent following product
Period: Overall Study
Arm/Group | ICD Patients (Single Arm Study)
Started | 504
Completed | 311
Not Completed | 193

BASELINE CHARACTERISTICS:
Arm/Group | ICD Patients
Number analyzed (Participants) | 504
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — data has been gathered based on information stored in the device. Data on sex is not available in this data.
  Male | NA — Data were not collected
Region of Enrollment [Number; unit: participants]
  Germany | 504

OUTCOME MEASURES:

1. Primary Outcome: Analysis of Change of Episodes Inappropriately Treated by Shock Therapy Due to Smart Shock™ Technology.
Description: Smart Shock technology is a suite of algorithms that are designed to prevent inappropriate shocks in ICD&CRT patients.
  Endpoints for the primary objective:
  * Episodes with shock therapy
  * Episodes without shock delivery due to Smart Shock™ technology
    * Episodes classified as supraventricular tachycardia (SVT) by PR Logic
    * Episodes classified as SVT by Wavelet
    * Shock therapy suppressed by T-wave Discrimination
    * Shock therapy suppressed by Lead Noise Discrimination
    * Shock therapy suppressed by Confirmation +
    * Episode with successful anti-tachycardia pacing (ATP) During Charging
Time Frame: 24 months
Population: The change of episodes of episodes inappropriately treated by shock due to Smart Shock™ was calculated as follow:
  change of episodes= (Episodes without shock therapy due to Smart Shock™)/(total number of episodes)
Measure: Number; unit: % of episodes wo shock due to SmartShock
Units Other Than Participants: total number of episodes
Groups:
- ICD Patients (Single Arm Study): Patients with an indication for an ICD implantation according to the guidelines treated with a Protecta™, Protecta™ XT or any equivalent following product
Arm/Group | ICD Patients (Single Arm Study)
Number analyzed (Participants) | 504
Number analyzed (total number of episodes) | 2529
% of episodes wo shock due to SmartShock | 94.9

2. Secondary Outcome: Number of Patients With All Smart Shock Algorithms Are Programmed on
Description: Endpoint: Patients, in which none of the Smart Shock algorithms is programmed "OFF" during the first Follow-Up after a maximum length of 90 days and 180 days.
Time Frame: 90 days or 180 days
Population: Patients with data available at 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | ICD Patients (Single Arm Study)
Number analyzed (Participants) | 427
Participants | 300

3. Secondary Outcome: Percentage of Patients, Without Shock Delivery Due to Smart Shock Technology
Description: Endpoint: Patients without shock delivery due to Smart Shock technology
Time Frame: 24 months
Measure: Number; unit: pat. w. at least 1 shock prevented in %
Arm/Group | ICD Patients (Single Arm Study)
Number analyzed (Participants) | 459
pat. w. at least 1 shock prevented in % | 15.3

4. Secondary Outcome: Analysis of the Number of Patients With Primary Preventive Indication for an ICD That Develop VF Episodes.
Description: Endpoint: Number of primary prevention patients with at least one ventricular fibrillation (VF) episode detected and successfully treated by the ICD
Time Frame: 24 months
Population: Of all 272 patients with primary preventive indication, only 265 patients had device data available for the Follow-Up period.
Measure: Count of Participants; unit: Participants
Arm/Group | ICD Patients
Number analyzed (Participants) | 265
Participants | 15

5. Secondary Outcome: Number of Patients That Developed AT/AF
Description: Endpoint: patients with >5 min atrial tachycardia/atrial fibrillation (AT/AF) in 'Daily Log' (Cardiac Compass)
Time Frame: 24 months
Population: Out of all patients analyzed (N=504), the patients with Single-Chamber-ICDs were excluded as these devices had no feature to identify AT/AF. This lead to N=367. Out of these 367 patients only 337 had Follow-Up data available whereas 30 patients only had implant data.
Measure: Count of Participants; unit: Participants
Arm/Group | ICD Patients (Single Arm Study)
Number analyzed (Participants) | 337
Participants | 117

6. Secondary Outcome: Analysis of the Proportion of Patients in Which ICD Parameters Remain on Nominal Programming.
Description: Endpoint: Deviation of ICD parameter programming in comparison to nominal programming at the first Follow-Up ≥ 90 days post-implant.
  Nominals for dual chamber ICD or cardiac resynchronization therapy (CRT) devices:
  * Lead Noise Discrimination = 'OnWithTimeout'
  * Lead Failure Predictor = 'On'
  * PR-Logic: AfibAflutter Rejection Rule = 'On'
  * PR-Logic: Sinus Tach Rejection Rule = 'On'
  * PR-Logic: Other 1:1 Rejection Rule = 'On'
  * High Rate Timeout = 'Off'
  * VF High Rate Timeout = 'Off'
  * Wavelet Rejection Rule = 'On'
  * VF Detection Interval = 320 and SVT Minimum Cycle Length = 260
  * T-Wave Oversensing Discrimination = 'On'
  * ATP During Charging = 'DuringCharging'
  Nominals for single chamber ICDs:
  * Lead Noise Discrimination = 'OnWithTimeout'
  * Lead Failure Predictor = 'On'
  * High Rate Timeout = 'Off'
  * VF High Rate Timeout = '0.75 min'
  * Wavelet Rejection Rule = 'On'
  * VF Detection Interval = 320 and SVT Minimum Cycle Length = 260
  * T-Wave Oversensing D
Time Frame: At the first Follow-Up ≥ 90 days post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | ICD Patients (Single Arm Study)
Number analyzed (Participants) | 427
Participants | 421

7. Secondary Outcome: Analysis of the Positive Predictive Value of the Investigated ICD Oversensing Algorithms
Description: Endpoint: Episode classified by the device as T-wave Oversensing or 'Noise'.
Time Frame: through study completion
Population: In total, 71 episodes were detected by the device and classified as T-wave Oversensing or Noise, but only 20 had electrogram (EGM) strips available. The analysis of the positive predictive value (PPV) was performed on these 20 episodes only. The number of true positives was 20. The number of false positives was 0.
Measure: Number; unit: Positive Predictive Value in %
Units Other Than Participants: episodes with EGM strips
Arm/Group | ICD Patients (Single Arm Study)
Number analyzed (Participants) | 4
Number analyzed (episodes with EGM strips) | 20
Positive Predictive Value in % | 100

ADVERSE EVENTS:
Time Frame: All devices that were used in this study are market-released and were only used within their approved indication. Therefore vigilance reporting was performed in the context of Post Market Surveillance. Adverse event information was therefore not collected during this study.
Description: All devices that were used in this study are market-released and were only used within their approved indication. Therefore vigilance reporting was performed in the context of Post Market Surveillance. Adverse event information was therefore not collected during this study.
Arm/Group | ICD Patients (Single Arm Study)
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
* No electronic case report form data available / only device data used
* Appropriateness of classification of Smart Shock algorithms not established; i.e. episode classification was limited to secondary endpoint 6
* No source data verification

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reviews publication within 3 weeks after submission of a manuscript. The sponsor can deny publication if the publication is not in accordance with the protocol, the publication would compromise business secrets or the issuing of patents or if the content of the publication is technically incorrect or may compromise other interests of the sponsor.